CLINICAL TRIAL: NCT02725567
Title: A Phase 3, 2 Part, Open-Label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Ivacaftor in Subjects With Cystic Fibrosis Who Are Less Than 24 Months of Age and Have an Ivacaftor-Responsive CFTR Mutation
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Ivacaftor in Subjects With Cystic Fibrosis Who Are Less Than 24 Months of Age and Have an Ivacaftor-Responsive CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX15-770-124; 2015-001997-16 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-04-01 (Estimated); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A: 3 to <24 months (Experimental): Participants weighing 5 to less than (<) 7 kilogram (kg) received 25 milligram (mg) IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA administered every 12 hours (q12h) on Days 1 through 3 and 1 morning dose on Day 4.
  Interventions: Drug: IVA
- Part B + A/B:1 to < 24 months (Experimental): Participants 4 to <6 months of age and weighing greater than or equal to (≥) 5 kg received 25 mg IVA q12h. At 6 months of age and older, participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h for 24 weeks on Part B. For Part A/B, participants 1 to <4 months weighing 3 kg to <5 kg received an initial low dose of 5.7 mg q12h IVA and those weighing ≥5 kg received 11.4 mg q12h IVA for the first 15 days of IVA treatment. Doses were maintained or adjusted upward at Day 15 and based on weight and/or age once they reached 4 months of age.
  Interventions: Drug: IVA

INTERVENTIONS:
Drug: IVA — Granules in sachet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
The purpose of this study was to evaluate the safety of ivacaftor treatment, and PK of ivacaftor and metabolites in participants with cystic fibrosis (CF) who are <24 months of age at treatment initiation and have an ivacaftor-responsive CF transmembrane conductance regulator (CFTR) gene mutation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF by sweat chloride value or CF mutation criteria.
* Have 1 of the following 10 CFTR mutations on at least 1 allele: G551D, G178R, S549N, S549R, G551S, G1244E, S1251N, S1255P, G1349D or R117H (eligible in regions where ivacaftor is approved for use). Part A/B group may also have other ivacaftor-responsive mutations.
* Hematology, serum chemistry, and vital signs results at screening with no clinically significant abnormalities that would interfere with the study assessments, as judged by the investigator.

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* Colonization with organisms associated with a more rapid decline in pulmonary status at screening (Only for Parts A and B)
* History of abnormal liver function or abnormal liver function at screening
* History of solid organ or hematological transplantation
* Use of any moderate or strong inducers or inhibitors of cytochrome P450 (CYP) 3A within 2 weeks before Day 1
* Participation in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 terminal half-lives before screening
* Hemoglobin (Hgb) <9.5 g/dL at screening
* Chronic kidney disease of Stage 3 or above
* Presence of a non-congenital or progressive lens opacity or cataract at Screening

Other protocol defined Inclusion/Exclusion Criteria may apply.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (13):
  - Birmingham, Alabama
  - Palo Alto, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (3):
  - Parkville, Victoria
  - South Brisbane
  - Westmead
- Toronto, Canada
- Dublin, Ireland
- United Kingdom (5):
  - Edinburgh
  - Leicester
  - London
  - Manchester
  - Oxford

REFERENCES:
- [Derived] Davies JC, Wainwright CE, Sawicki GS, Higgins MN, Campbell D, Harris C, Panorchan P, Haseltine E, Tian S, Rosenfeld M. Ivacaftor in Infants Aged 4 to <12 Months with Cystic Fibrosis and a Gating Mutation. Results of a Two-Part Phase 3 Clinical Trial. Am J Respir Crit Care Med. 2021 Mar 1;203(5):585-593. doi: 10.1164/rccm.202008-3177OC. PMID 33023304
- [Derived] Rosenfeld M, Wainwright CE, Higgins M, Wang LT, McKee C, Campbell D, Tian S, Schneider J, Cunningham S, Davies JC; ARRIVAL study group. Ivacaftor treatment of cystic fibrosis in children aged 12 to <24 months and with a CFTR gating mutation (ARRIVAL): a phase 3 single-arm study. Lancet Respir Med. 2018 Jul;6(7):545-553. doi: 10.1016/S2213-2600(18)30202-9. Epub 2018 Jun 7. PMID 29886024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in participants with cystic fibrosis (CF) who were less than (<) 24 months of age at Day 1 and have an ivacaftor-responsive CF transmembrane conductance regulator (CFTR) mutation.
Groups:
- Part A: 3 to < 24 Months: Participants weighing 5 to less than (<) 7 kilogram (kg) received 25 milligram (mg) IVA (ivacaftor), 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA administered every 12 hours (q12h) on Days 1 through 3 and 1 morning dose on Day 4.
- Part B + A/B: 1 to < 24 Months: Participants 4 to <6 months of age and weighing greater than or equal to (≥) 5 kg received 25 mg IVA q12h. At 6 months of age and older, participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h for 24 weeks on Part B.
  For Part A/B, participants 1 to <4 months weighing 3 kg to <5 kg received an initial low dose of 5.7 mg q12h IVA and those weighing ≥5 kg received 11.4 mg q12h IVA for the first 15 days of IVA treatment. Doses were maintained or adjusted upward at Day 15 and based on weight and/or age once they reached 4 months of age.
Period: Part A (Up to 5 Days)
Arm/Group | Part A: 3 to < 24 Months | Part B + A/B: 1 to < 24 Months
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0
Period: Part B + A/B ( Up to 24 Weeks)
Arm/Group | Part A: 3 to < 24 Months | Part B + A/B: 1 to < 24 Months
Started | 0 | 43 (Out of the 19 participants in the reporting arm Part A, 5 also participated in the reporting arm "Part B + Part A/B.)
Completed | 0 | 40
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal of Consent (not due to adverse event) | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Groups:
- Ivacaftor (IVA): Part A: Participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA administered q12h on Days 1 through 3 and 1 morning dose on Day 4.
  Participants 4 to <6 months of age and ≥5 kg received 25 mg IVA q12h. At 6 months of age and older, participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h for 24 weeks on Part B.
  For Part A/B, participants 1 to <4 months weighing 3 kg to <5 kg received an initial low dose of 5.7 mg q12h IVA and those weighing ≥5 kg received 11.4 mg q12h IVA for the first 15 days of IVA treatment. Doses were maintained or adjusted upward at Day 15 and based on weight and/or age once they reached 4 months of age.
Arm/Group | Ivacaftor (IVA)
Number analyzed (Participants) | 57
Age, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and for the combined Part B+ A/B. Here, "Number Analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 19
    Part A: 12 to <24 months | 7
    Part A: 6 to <12 months | 6
    Part A: 4 to <6 months | 4
    Part A: 1 to <4 months | 2
    Part B+ A/B: number analyzed (Participants) | 43
    Part B+ A/B: 12 to <24 months | 19
    Part B+ A/B: 6 to <12 months | 11
    Part B+ A/B: 4 to <6 months | 6
    Part B+ A/B: 1 to <4 months | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and for the combined Part B+ A/B. Here, "Number Analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 19
    Part A: Female | 10
    Part A: Male | 9
    Part B + A/B: number analyzed (Participants) | 43
    Part B + A/B: Female | 22
    Part B + A/B: Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and for the combined Part B+ A/B. Here, "Number Analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 19
    Part A: Hispanic or Latino | 0
    Part A: Not Hispanic or Latino | 19
    Part A: Not collected per local regulations | 0
    Part B + A/B: number analyzed (Participants) | 43
    Part B + A/B: Hispanic or Latino | 1
    Part B + A/B: Not Hispanic or Latino | 42
    Part B + A/B: Not collected per local regulations | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A and for the combined Part B+ A/B. Here, "Number Analyzed" signifies participants who were evaluable for specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 19
    Part A: White | 19
    Part A: Black or African American | 0
    Part A: Asian | 0
    Part A: American Indian or Alaska Native | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0
    Part A: Not collected per local Regulations | 0
    Part B + A/B: number analyzed (Participants) | 43
    Part B + A/B: White | 43
    Part B + A/B: Black or African American | 0
    Part B + A/B: Asian | 0
    Part B + A/B: American Indian or Alaska Native | 0
    Part B + A/B: Native Hawaiian or Other Pacific Islander | 0
    Part B + A/B: Not collected per local Regulations | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious (TEAEs)
Time Frame: Day 1 through Day 70
Population: Safety set included all participants who received at least 1 dose of study drug in Part A. This outcome measure was planned only for Part A: 3 to <24 months arm.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: 3 to < 24 Months: Participants weighing 5 to <7 kg received 25 mg IVA, weighing 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h on Days 1 through Day 3 and 1 morning dose on Day 4.
Arm/Group | Part A: 3 to < 24 Months
Number analyzed (Participants) | 19
Participants
  Participants with TEAEs | 10
  Participants with Serious TEAEs | 1

2. Primary Outcome: Part A: Observed Plasma Concentration of IVA and Their Metabolites (M1-IVA and M6-IVA)
Time Frame: Pre-dose, 2-4 hours, 6-8 hours, 24-60 hours post-dose
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug in Part A. Here the "Number Analyzed" signifies those participants who were evaluable for the specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Part A: 3 to < 24 Months
Number analyzed (Participants) | 19
nanogram per milliliter (ng/ml)
  Pre dose: IVA | 654 (531)
  Pre dose: M1-IVA | 1880 (1160)
  Pre dose: M6-IVA | 2680 (1990)
  2-4 hrs post dose: IVA | 956 (497)
  2-4 hrs post dose: M1-IVA | 1990 (1160)
  2-4 hrs post dose: M6-IVA | 2460 (2110)
  6-8 hrs post dose: IVA | 1040 (623)
  6-8 hrs post dose: M1-IVA | 2440 (1260)
  6-8 hrs post dose: M6-IVA | 2880 (2180)
  24-60 hrs post dose: IVA: number analyzed (Participants) | 18
  24-60 hrs post dose: IVA | 129 (68.8)
  24-60 hrs post dose: M1-IVA: number analyzed (Participants) | 18
  24-60 hrs post dose: M1-IVA | 508 (228)
  24-60 hrs post dose: M6-IVA: number analyzed (Participants) | 18
  24-60 hrs post dose: M6-IVA | 1100 (982)

3. Primary Outcome: Part B +A/B: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious (TEAEs)
Time Frame: Day 1 through Week 38
Population: Safety Set included all participants who received at least 1 dose of study drug. The safety and tolerability analyses were assessed for the overall treatment arm. Therefore, the analysis is reported in a overall Part B+ A/B: 1 to <24 months arm.
Measure: Count of Participants; unit: Participants
Groups:
- Part B + A/B: 1 to <24 Months: Participants 4 to <6 months of age and ≥5 kg received 25 mg IVA q12h. At 6 months of age and older, participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h for 24 weeks on Part B.
  For Part A/B, participants 1 to <4 months weighing 3 kg to <5 kg received an initial low dose of 5.7 mg q12h IVA and those weighing ≥5 kg received 11.4 mg q12h IVA for the first 15 days of IVA treatment. Doses were maintained or adjusted upward at Day 15 and based on weight and/or age once they reached 4 months of age.
Arm/Group | Part B + A/B: 1 to <24 Months
Number analyzed (Participants) | 43
Participants
  Participants with TEAEs | 38
  Participants with Serious (TEAEs) | 6

4. Primary Outcome: Part A/B: Observed Plasma Concentration of IVA and Their Metabolites (M1-IVA and M6-IVA)
Time Frame: Day 4 (pre-dose, 2-4 hours, 6-8 hours post-dose); Day 15 (pre-dose); Week 4 (pre-dose); Week 8 (pre-dose, 2-4 hours, 6-8 hours post-dose); Week 12 (pre-dose); Week 18 (pre-dose) and Week 24 (pre-dose)
Population: PK set included participants who received at least 1 dose of study drug in Part A/B. Here the "Number Analyzed" signifies those participants who were evaluable for the specified time point.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Part A/B: 1 to <4 Months: Participants 1 to <4 months weighing 3 kg to <5 kg received an initial low dose of 5.7 mg q12h IVA and those weighing ≥5 kg received 11.4 mg q12h IVA for the first 15 days of IVA treatment. Doses were maintained or adjusted upward at Day 15 and based on weight and/or age once they reached 4 months of age.
Arm/Group | Part A/B: 1 to <4 Months
Number analyzed (Participants) | 7
ng/ml
  Day 4 (pre dose): IVA | 348 (151)
  Day 4 (pre dose): M1-IVA | 867 (412)
  Day 4 (pre dose): M6-IVA | 1570 (570)
  Day 4 (2-4 hrs post dose): IVA | 381 (135)
  Day 4 (2-4 hrs post dose): M1-IVA | 851 (333)
  Day 4 (2-4 hrs post dose): M6-IVA | 1370 (450)
  Day 4 (6-8 hrs post dose): IVA | 501 (196)
  Day 4 (6-8 hrs post dose): M1-IVA | 1190 (420)
  Day 4 (6-8 hrs post dose): M6-IVA | 1670 (551)
  Day 15 (pre dose): IVA: number analyzed (Participants) | 6
  Day 15 (pre dose): IVA | 191 (134)
  Day 15 (pre dose): M1-IVA: number analyzed (Participants) | 6
  Day 15 (pre dose): M1-IVA | 614 (378)
  Day 15 (pre dose): M6-IVA: number analyzed (Participants) | 6
  Day 15 (pre dose): M6-IVA | 1510 (1110)
  Week 4 (pre dose): IVA: number analyzed (Participants) | 6
  Week 4 (pre dose): IVA | 316 (130)
  Week 4 (pre dose): M1-IVA: number analyzed (Participants) | 6
  Week 4 (pre dose): M1-IVA | 1170 (577)
  Week 4 (pre dose): M6-IVA: number analyzed (Participants) | 6
  Week 4 (pre dose): M6-IVA | 3370 (2330)
  Week 8 (pre dose): IVA | 449 (352)
  Week 8 (pre dose): M1-IVA | 1030 (476)
  Week 8 (pre dose): M6-IVA | 2380 (1500)
  Week 8 (2-4 hrs post dose): IVA | 523 (262)
  Week 8 (2-4 hrs post dose): M1-IVA | 1360 (982)
  Week 8 (2-4 hrs post dose): M6-IVA | 2100 (1540)
  Week 8 (6-8 hrs post dose): IVA | 438 (79.8)
  Week 8 (6-8 hrs post dose): M1-IVA | 1420 (606)
  Week 8 (6-8 hrs post dose): M6-IVA | 2320 (1330)
  Week 12 (pre dose): IVA: number analyzed (Participants) | 5
  Week 12 (pre dose): IVA | 213 (173)
  Week 12 (pre dose): M1-IVA: number analyzed (Participants) | 5
  Week 12 (pre dose): M1-IVA | 906 (660)
  Week 12 (pre dose): M6-IVA: number analyzed (Participants) | 5
  Week 12 (pre dose): M6-IVA | 2500 (1760)
  Week 18 (pre dose): IVA: number analyzed (Participants) | 6
  Week 18 (pre dose): IVA | 226 (153)
  Week 18 (pre dose): M1-IVA: number analyzed (Participants) | 6
  Week 18 (pre dose): M1-IVA | 815 (470)
  Week 18 (pre dose): M6-IVA: number analyzed (Participants) | 6
  Week 18 (pre dose): M6-IVA | 2060 (1190)
  Week 24 (pre dose): IVA: number analyzed (Participants) | 6
  Week 24 (pre dose): IVA | 276 (137)
  Week 24 (pre dose): M1-IVA: number analyzed (Participants) | 6
  Week 24 (pre dose): M1-IVA | 1120 (496)
  Week 24 (pre dose): M6-IVA: number analyzed (Participants) | 6
  Week 24 (pre dose): M6-IVA | 2380 (799)

5. Secondary Outcome: Part B: Observed Plasma Concentration of IVA and Their Metabolites (M1-IVA and M6-IVA)
Time Frame: Week 2 (pre-dose, 2-4 hours, 6-8 hours post-dose); Week 8 (pre-dose,1 hour, 4-hour post-dose); Week 24 (pre-dose, 2-4 hours post dose)
Population: PK set included participants who received at least 1 dose of study drug in Part B. Here the "Number Analyzed" signifies those participants who were evaluable for the specified time point.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Part B: 4 to <24 Months: Participants 4 to <6 months of age and ≥5 kg received 25 mg IVA q12h. At 6 months of age and older, participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h for 24 weeks on Part B.
Arm/Group | Part B: 4 to <24 Months
Number analyzed (Participants) | 35
ng/ml
  Week 2 (pre dose): IVA: number analyzed (Participants) | 34
  Week 2 (pre dose): IVA | 457 (441)
  Week 2 (pre dose): M1-IVA: number analyzed (Participants) | 34
  Week 2 (pre dose): M1-IVA | 1340 (934)
  Week 2 (pre dose): M6-IVA: number analyzed (Participants) | 34
  Week 2 (pre dose): M6-IVA | 1980 (1790)
  Week 2 (2-4 hrs post dose): IVA: number analyzed (Participants) | 34
  Week 2 (2-4 hrs post dose): IVA | 812 (726)
  Week 2 (2-4 hrs post dose): M1-IVA: number analyzed (Participants) | 34
  Week 2 (2-4 hrs post dose): M1-IVA | 1560 (1190)
  Week 2 (2-4 hrs post dose): M6-IVA: number analyzed (Participants) | 34
  Week 2 (2-4 hrs post dose): M6-IVA | 1770 (1970)
  Week 2 (6-8 hrs post dose): IVA: number analyzed (Participants) | 32
  Week 2 (6-8 hrs post dose): IVA | 969 (705)
  Week 2 (6-8 hrs post dose): M1-IVA: number analyzed (Participants) | 32
  Week 2 (6-8 hrs post dose): M1-IVA | 2210 (1360)
  Week 2 (6-8 hrs post dose): M6-IVA: number analyzed (Participants) | 32
  Week 2 (6-8 hrs post dose): M6-IVA | 2140 (1880)
  Week 8 (pre dose): IVA: number analyzed (Participants) | 34
  Week 8 (pre dose): IVA | 404 (376)
  Week 8 (pre dose): M1-IVA: number analyzed (Participants) | 34
  Week 8 (pre dose): M1-IVA | 1220 (782)
  Week 8 (pre dose): M6-IVA: number analyzed (Participants) | 34
  Week 8 (pre dose): M6-IVA | 1720 (1110)
  Week 8 (1 hrs post dose): IVA: number analyzed (Participants) | 33
  Week 8 (1 hrs post dose): IVA | 466 (384)
  Week 8 (1 hrs post dose): M1-IVA: number analyzed (Participants) | 33
  Week 8 (1 hrs post dose): M1-IVA | 1100 (670)
  Week 8 (1 hrs post dose): M6-IVA: number analyzed (Participants) | 33
  Week 8 (1 hrs post dose): M6-IVA | 1500 (881)
  Week 8 (4 hrs post dose): IVA: number analyzed (Participants) | 33
  Week 8 (4 hrs post dose): IVA | 996 (520)
  Week 8 (4 hrs post dose): M1-IVA: number analyzed (Participants) | 33
  Week 8 (4 hrs post dose): M1-IVA | 2130 (950)
  Week 8 (4 hrs post dose): M6-IVA: number analyzed (Participants) | 33
  Week 8 (4 hrs post dose): M6-IVA | 1750 (1010)
  Week 24 (pre dose): IVA | 301 (204)
  Week 24 (pre dose): M1-IVA | 1050 (492)
  Week 24 (pre dose): M6-IVA | 1600 (783)
  Week 24 (2-4 hrs post dose): IVA: number analyzed (Participants) | 34
  Week 24 (2-4 hrs post dose): IVA | 794 (480)
  Week 24 (2-4 hrs post dose): M1-IVA: number analyzed (Participants) | 34
  Week 24 (2-4 hrs post dose): M1-IVA | 1540 (783)
  Week 24 (2-4 hrs post dose): M6-IVA: number analyzed (Participants) | 34
  Week 24 (2-4 hrs post dose): M6-IVA | 1320 (592)

6. Secondary Outcome: Part B + A/B: Absolute Change From Baseline in Sweat Chloride
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 24
Population: The Full Analysis Set (FAS) included all enrolled participants who were exposed to any amount of study drug in Part B + A/B. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Groups:
- Part B + A/B: 1 to < 24 Months: Participants 4 to <6 months of age and ≥5 kg received 25 mg IVA q12h. At 6 months of age and older, participants weighing 5 to <7 kg received 25 mg IVA, 7 to <14 kg received 50 mg IVA, and those weighing 14 to <25 kg received 75 mg IVA q12h for 24 weeks on Part B.
  For Part A/B, participants 1 to <4 months weighing 3 kg to <5 kg received an initial low dose of 5.7 mg q12h IVA and those weighing ≥5 kg received 11.4 mg q12h IVA for the first 15 days of IVA treatment. Doses were maintained or adjusted upward at Day 15 and based on weight and/or age once they reached 4 months of age.
Arm/Group | Part B + A/B: 1 to < 24 Months
Number analyzed (Participants) | 23
millimole per liter (mmol/L) | -62.0 (22.2)

ADVERSE EVENTS:
Time Frame: From Day 1 Through Safety Follow-up Period (up to Day 70 for Part A and up to Week 38 for Part B + A/B)
Groups:
- Part A: 3 to < 24 Months: Participants weighing 5 to <7 kg received 25 mg IVA, weighing 7 to <14 kg received 50 mg IVA, and participants weighing 14 to < 25 kg received 75 mg IVA q12h on days 1 through day 3 and 1 morning dose on day 4.
Arm/Group | Part A: 3 to < 24 Months | Part B + A/B: 1 to <24 Months
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/19 | 6/43
Other Adverse Events (participants affected / at risk) | 10/19 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 3 to < 24 Months (N=19) | Part B + A/B: 1 to <24 Months (N=43)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Eczema Coxsackium (Infections and infestations) | 0 | 1
Eczema herpeticum (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 3 to < 24 Months (N=19) | Part B + A/B: 1 to <24 Months (N=43)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Infantile spitting up (Gastrointestinal disorders) | 1 | 0
Teething (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 8
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 12
Ear infection (Infections and infestations) | 0 | 3
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 3
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 7
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 7
Blood pressure increased (Investigations) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
Pseudomonas test positive (Investigations) | 0 | 3
Sleep disorder (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 24
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 2
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02725567/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT02725567/SAP_001.pdf